CLINICAL TRIAL: NCT04353700
Title: Does a 12-week Home-based Dynamic Yoga Intervention Improve Bone and Cardiovascular Health in Healthy Premenopausal Women? A Randomized Controlled Feasibility Study
Brief Title: Effects of a 12-week Home-based Yoga on Bone and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Lowell (Other)
Responsible Party: Principal Investigator, SoJung Kim, Assistant Professor, University of Massachusetts, Lowell
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-183-KIM-XPD
Record Dates: First submitted 2020-04-10; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Osteoporosis; Cardiovascular Risk Factor
Keywords: Yoga; Bone markers; Arterial stiffness; Premenopausal women
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned either a yoga intervention group or a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga group (Active Comparator): A certified yoga instructor led the supervised yoga session. An exercise physiologist taught how to record your Rating of Perceived Exertion to monitor their exercise intensity during the in-home yoga intervention. During the in-home yoga intervention, participants performed 30 to 50 minutes of yoga postures three to five times a week for 12 weeks.
  Interventions: Behavioral: Yoga group
- Control group (No Intervention): If participants were in a CON group, they did not receive the yoga intervention. Instead, they were encouraged to maintain a normal daily lifestyle monitored by the BPAQ at one-month intervals during the 12-week intervention.

INTERVENTIONS:
Behavioral: Yoga group — During the in-home yoga intervention, participants performed 30 to 50 minutes of yoga postures three to five times a week for 12 weeks, including 5 minutes of warm-up exercise, 15 to 30 minutes of dynamic flow yoga postures, 10 minutes of weight barring standing postures, and 5 minutes of cool-down. These in-home sessions were a repeat of what participants learned during the first week of training session at UML. We progressively increased the intensity of the home practice sessions by adding the number of sun salutation (SS) over the 12 weeks.
  Arms: Yoga group

SUMMARY:
While effects of specific exercise interventions on bone and CVD in postmenopausal women have been demonstrated and evaluated, the effects of randomized controlled exercise interventions, particularly in middle-aged premenopausal women are sparse. Therefore, it is imperative to examine the relation between behavioral interventions and bone and cardiovascular outcomes in premenopausal women as this understudied group is at high risk for the initial stages of bone loss and cardiovascular disease development.

DETAILED DESCRIPTION:
Presently, it is not clear whether the intensity of Yoga interventions is high enough to induce positive effects on bone and cardiovascular health in a healthy population. For example, Hagins et al. (2007) reported that the metabolic costs of Hatha Yoga, averaged across the entire session, represent low levels of physical activity (walking). On the other hand, Ashtanga Yoga, or power Yoga, is performed at a higher intensity than Hatha Yoga and has been shown to elicit significantly higher heart rates than either Hatha or gentle Yoga (Cowen and Adams, 2007). Sun Salutations (SS) are an example of an Ashtanga Yoga sequence, where yoga postures are performed dynamically with combinations of forward and backward bending poses (Omkar et al., 2011). A previous 8-month yoga intervention found that regular long-term Ashtanga yoga had a small positive effect on bone formation in premenopausal women. Although Yoga has the potential to be an alternative physical activity to improve bone health and arterial stiffness, there is a lack of high-quality evidence for this type of intervention. Thus, the purpose of this study is to assess the feasibility of a 12-week home-based dynamic yoga intervention designed to improve bone metabolism and arterial stiffness in healthy premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Participants were healthy premenopausal women volunteers between the ages of 30 and 48 years.
* Participants were free of chronic back or joint problems, cardiovascular disease, non-smokers, not pregnant, not taking antihypertensive drugs or any medication that affects bone density.
* Participants didn't have regularly participated in a weight training program and yoga exercise at least 12 months prior to the study.
* Participants were medically stable, ambulatory, and capable of training.

Exclusion Criteria:

* Individual who were outside of the 30-48 years age range and who exceed the weight limit of the DXA (300 pounds).
* Individuals who did not have the regular menstrual cycles.
* Pregnancy or the possibility of becoming pregnant during the intervention period
* Individuals who were taking medications known to affect bone metabolism such as steroid hormones, calcitonin, or corticosteroids.
* Any persons with physical and mental disabilities preventing them from being trained, including orthopedic or arthritic problems, were not allowed to participate.
* Individuals whose radiation exposure from medical and/or research tests in the previous year exceeds the recommended regulator limit.

Ages: 30 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females who have regular menstrual cycles
Enrollment: 35 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity participation was assessed. | BPAQ scores were collected at baseline, at 6 weeks, and after 12 weeks to see any differences throughout the intervention periods.
  Participants were asked to fill out a physical activity questionnaire (BPAQ scores) Physical activity participation was estimated with the bone-specific physical activity questionnaire (BPAQ score).
Change in Health history was assessed. | HH questionnaires were collected at baseline, at 6 weeks, and after 12 weeks to see any changes throughout the intervention periods.
  A health history questionnaire (HH) was utilized to examine any medical history that can affect bone and cardiovascular health.
Change in menstrual history was assessed | MH questionnaires were collected at baseline, at 6 weeks, and after 12 weeks to see any changes throughout the intervention periods.
  A menstrual history questionnaire (MH) was used to determine if a participant was pregnant.
Change in calcium intake was assessed | CI questionnaires were collected at baseline, at 6 weeks, and after 12 weeks to see any changes throughout the intervention periods.
  Daily calcium intake (mg/d) was estimated using a calcium intake questionnaire (CI).
Change in Body Mass Index (BMI) was assessed | Height and weight were collected at baseline and after 12 weeks.
  Height (cm) and weight (kg) were collected to calculate BMI (kg/m2).
Change in total fat mass was assessed | Total fat mass was measured at baseline and after 12 weeks.
  Total fat mass (g) was measured using Dual Energy-X-ray Absorptiometry.
Change in bone free lean body mass was assessed | Bone free lean body mass was measured at baseline and after 12 weeks.
  Bone free lean body mass (g) was measured using Dual Energy-X-ray Absorptiometry.
Change in %fat was assessed | %fat was measured at baseline and after 12 weeks.
  %fat (%) was measured using Dual Energy-X-ray Absorptiometry.
Change in P1NP was assessed. | Blood draws were collected at baseline, at 6 weeks, and after 12 weeks.
  A blood draw (approximately 10 ml) was collected to investigate differences in bone formation marker (P1NP, ng/mL)
Change in CTX was assessed | Blood draws were collected at baseline, at 6 weeks, and after 12 weeks.
  A blood draw (approximately 10 ml) was collected to investigate differences in bone resorption marker (CTX, ng/mL)

SECONDARY OUTCOMES:
Change in Arterial stiffness was assessed | Arterial stiffness was collected at baseline, at 6 weeks, and after 12 weeks
  Arterial stiffness (m/s) was measured using Pulse Wave Velocity (PWV) to look at intervention effects.

CONTACTS AND LOCATIONS:
Overall Officials: SoJung Kim, PhD, Principal Investigator — University of Massachusetts, Lowell
Locations (1):
- University of Massachusetts, Lowell, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No